CLINICAL TRIAL: NCT02389114
Title: Effect of Soy Protein and Polydextrose on Food Intake in Young Chinese Adult Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 2013/00383
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Satiety; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Soybean Proteins; polydextrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Protein Preload (Active Comparator): The subjects consumed soybean curd preload containing low protein content.
  Interventions: Other: Soy Protein
- Low Protein with Polydextrose Preload (Experimental): The subjects consumed soybean curd preload containing low protein content and polydextrose.
  Interventions: Other: Soy Protein; Other: Polydextrose
- High Protein Preload (Experimental): The subjects consumed soybean curd preload containing high protein content.
  Interventions: Other: Soy Protein
- High Protein with Polydextrose Preload (Experimental): The subjects consumed soybean curd preload containing high protein content and polydextrose.
  Interventions: Other: Soy Protein; Other: Polydextrose

INTERVENTIONS:
Other: Soy Protein — Soy protein is commonly consumed in Asian diet.
Other: Polydextrose — Polydextrose is a randomly bonded polymer of glucose developed in the 1960s. It is widely recognized as a soluble fiber that is not digested in the upper gastrointestinal tract due to the complex structure and nature of the glycosidic bonds, but is partially fermented by the microbiota in large intestine generating short chain fatty acids.
  Other Names: Litesse
  Arms: High Protein with Polydextrose Preload; Low Protein with Polydextrose Preload

SUMMARY:
The primary hypothesis of this study is that the higher concentration of soy protein intake will increase satiety and decrease the energy intake at the subsequent meal.

The secondary hypothesis is that the synergistic effect of soy protein and polydextrose will further increase satiety and reduce energy intake at the subsequent meal.

The third hypothesis is that the ingestion of protein and polydextrose will differentially impact on satiety-related metabolism, i.e. blood glucose, insulin, urea, plasma amino acids, gut hormones and gastric emptying.

DETAILED DESCRIPTION:
Soy foods have been part of Asian food systems for millennia. In the past decades, both soy proteins and polydextrose have been widely used in a variety of food products. Helping consumers to feel less hungry is an approach to weight management because it has the potential to decrease inter-meal hunger and hence reduce overall energy intake. Considering the possible satiety effect of soy protein and polydextrose, inclusion of these molecules in the diet could therefore potentially reduce the energy intake and assist with weight management in order to attenuate the rise in obesity incidence globally. The study will provide data for the first time on how soy protein and soluble fiber impact on satiety and acute energy intake in those of Chinese ethnic origin. The research sets out to determine the effect of soy protein and polydextrose on satiety and food intake in Asians. It specifically attempts to comprehend the physiological mechanisms involving blood glucose, insulin, urea, plasma amino acids, gut hormones and the rate of gastric emptying of soy protein and polydextrose on appetite ratings, satiety and subsequent food intake. The study will recruit healthy young Chinese male, who will return for four test sessions on non-consecutive days. At each session, the subjects will be given a standard breakfast, followed 180 min later by a soybean curd preload and a buffet lunch 90 min after the preload. Four preloads will be tested: (1) low protein, (2) high protein, (3) low protein with polydextrose, and (4) high protein with polydextrose. Each soybean curd preload will be tested once by each subject. Blood samples from cannulated veins and fingerpricks will be collected before the preload, 15, 30, 45, 60, 75 and 90 min after the preload for the analysis of glucose, insulin, urea, plasma amino acids, and gut hormones. At the same time points as when blood samples collected, gastric emptying measurements will be carried out using ultrasound. Subjective motivational ratings for hunger, fullness, desire to eat and prospective food consumption will be measured by the use of visual analogue scales (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Males
* Chinese ethnicity
* Age between 21-40 years
* Body mass index (BMI) between 18-24 kg/m2
* Healthy
* Normal blood pressure (120/80 mm Hg)
* Fasting blood glucose < 6 mmol/L

Exclusion Criteria:

* Having eating disorders or conscious restriction of food intake
* Partaking in sports at the competitive and endurance levelsHaving allergies/ intolerances to the foods presented in the study
* Having metabolic diseases (diabetes, hypertension and the metabolic syndrome) or chronic gastrointestinal disorders
* Having regime diets (for medical or aesthetic reasons)
* Having medical conditions requiring prescription medication and taking medications known to affect appetite (steroids, sulphonylureas, antihistamines, antidepressants, amphetamines, hypoglycaemic agents and hormones).
* Smoking

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Food intake | 90 min subsequent to preload consumption
  Ad-libitum lunch will be provided to measure food intake

SECONDARY OUTCOMES:
Subjective motivational ratings | VAS will be obtained before and after breakfast, 1 and 2 h after breakfast, before preload, 15, 30, 45, 60, and 75 min after the preload, and before and after lunch.
  Subjective motivational ratings for hunger, fullness, desire to eat and prospective food consumption was measured by the use of visual analogue scales (VAS).
Gastric emptying rate | Before the preload, and 15, 30, 45, 60, 75 and 90 min after the preload
  The rate of gastric emptying was measured by the use of ultrasound scanning.
Physiological Outcomes | Before the preload, and 15, 30, 45, 60, 75 and 90 min after the preload
  Blood samples were obtained to analyze glucose, insulin, plasma amino acids, and gut hormones gut hormones